CLINICAL TRIAL: NCT00592163
Title: Phase I Study of Oral ZIO-101-C in Advanced Solid Tumors and Lymphomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGC1002
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Solid Tumors; Lymphomas
Keywords: Cancer; Arsenic
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — darinaparsin

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ZIO-101-C (Darinaparsin)

INTERVENTIONS:
Drug: ZIO-101-C (Darinaparsin) — Dose Escalation study, 200 mg - 900 mg, cumulative daily dose split to be taken BID 7 times a week (>8 hours between doses) for 3 weeks followed by 1 week of rest
  Other Names: ZIO-101-C

SUMMARY:
A Phase I Study of Oral ZIO-101-C in Advanced Solid Tumors and Lymphomas

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histological or cytological confirmation of advanced cancer that is refractory to standard therapies for their condition.
2. Men and women of ≥18 years of age.
3. ECOG performance score ≤2.
4. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions MUST NOT have been in a previously irradiated field or injected with biological agents. Eligible subjects with lymphomas must have measurable disease as defined by the revised International Working Group response criteria.
5. Life expectancy ≥12 weeks.
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements, to be conducted <2 weeks prior to Baseline:

   * Creatinine ≤1.5 × upper limit of normal (ULN) OR a calculated creatinine clearance ≥50 cc/min
   * Total bilirubin ≤2 × ULN
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤3 × ULN
   * Granulocytes in peripheral blood ≥1 × 109/L, hemoglobin ≥10 g/dL, and platelets ≥50,000 /μL
7. Adequate vascular access for repeated blood sampling.
8. Men and women of childbearing potential must agree to use effective contraception from Screening through the duration of Study participation.
9. Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee (IEC/IRB) having jurisdiction over the site.

Exclusion Criteria:

1. New York Heart Association (NYHA) functional class ≥3 myocardial infarction within 6 months
2. Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; a QTc ≥450 msec; or a ≥Grade 2 atrioventricular (AV) block or left bundle branch block (LBBB); or documented history of prolonged QTc.
3. Pregnant and/or lactating women.
4. Uncontrolled systemic infection (documented with microbiological studies).
5. Metastatic brain or meningeal tumors.
6. Subjects with seizure disorder requiring medication (such as anti-epileptics).
7. History of confusion or dementia or neurological condition that could mask a potential adverse response to the Study Drug, which may include transient ischemic attack, Parkinson's disease, thrombotic or hemorrhagic stroke, Alzheimers, and other neurological disorders.
8. Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of Study entry (mitomycin C or nitrosureas should not be given within 6 weeks of Study entry).
9. Radiotherapy during study or within 3 weeks of Study entry.
10. Surgery within 4 weeks of start of Study Drug dosing.
11. Investigational drug therapy outside of this trial during or within 4 weeks of Study entry.
12. History of invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
13. Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the study or evaluation of Study results.
14. Any condition that is unstable or could jeopardize the safety of the subject and his/her compliance in the Study.
15. Arsenic allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-12; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal, Quebec, Canada